CLINICAL TRIAL: NCT07061704
Title: Oncolytic Virus Combined With Chemotherapy and Immune Checkpoint Inhibitors in Patients With Initially Unresectable Locally Advanced Esophageal Squamous Cell Carcinoma：An Open-label, Single-arm Phase II Study
Brief Title: Oncolytic Virus in Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Clinical Professor, Sichuan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VOLCAN-251
Record Dates: First submitted 2025-06-29; First posted 2025-07-11 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; Oncolytic Virus; clinical efficacy; safety; Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oncolytic virus + chemotherapy + PD-1 inhibitor (Experimental): Oncolytic Virus: Administered via intratumoral (metastatic lesions in the neck or supraclavicular lymph nodes) injection once every 3 weeks, for a total of two doses, or until disease progression, the occurrence of unacceptable toxicity, or death from any cause, whichever occurs first.Chemotherapy + Immune Checkpoint Inhibitor (ICI): Administered via intravenous infusion once every 3 weeks.
  Interventions: Biological: Oncolytic Virus: Administered via intratumoral injection (metastatic lesions in the neck or supraclavicular lymph nodes) once every 3 weeks, for a total of two to four doses.
- Oncolytic virus in primary lesion + chemotherapy + PD-1 inhibitor (Experimental): Oncolytic Virus: Administered via intratumoral (primary lesion of ESCC) injection once every 3 weeks, for a total of two doses, or until disease progression, the occurrence of unacceptable toxicity, or death from any cause, whichever occurs first.Chemotherapy + Immune Checkpoint Inhibitor (ICI): Administered via intravenous infusion once every 3 weeks.
  Interventions: Biological: Oncolytic Virus: Administered via intratumoral injection (primary lesions) once every 3 weeks, for a total of two to four doses.

INTERVENTIONS:
Biological: Oncolytic Virus: Administered via intratumoral injection (metastatic lesions in the neck or supraclavicular lymph nodes) once every 3 weeks, for a total of two to four doses. — Oncolytic Virus: Administered via intratumoral injection(metastatic lesions in the neck or supraclavicular lymph nodes) once every 3 weeks, for a total of two to four doses, or until disease progression, the occurrence of unacceptable toxicity, or death from any cause, whichever occurs first. Chemotherapy + Immune Checkpoint Inhibitor (ICI): Administered via intravenous infusion once every 3 weeks.
  Arms: Oncolytic virus + chemotherapy + PD-1 inhibitor
Biological: Oncolytic Virus: Administered via intratumoral injection (primary lesions) once every 3 weeks, for a total of two to four doses. — Oncolytic Virus: Administered via intratumoral injection (primary lesions) once every 3 weeks, for a total of two to four doses, , or until disease progression, the occurrence of unacceptable toxicity, or death from any cause, whichever occurs first. Chemotherapy + Immune Checkpoint Inhibitor (ICI): Administered via intravenous infusion once every 3 weeks.
  Arms: Oncolytic virus in primary lesion + chemotherapy + PD-1 inhibitor

SUMMARY:
This clinical trial is designed to evaluate the preliminary efficacy and safety of an oncolytic virus combined with chemotherapy and an immune checkpoint inhibitor in patients with initially unresectable, locally advanced esophageal squamous cell carcinoma (ESCC). The primary endpoints are safety, surgical conversion rate and event-free survival (EFS). Secondary endpoints include overall survival (OS), objective response rate (ORR), and quality of life (QoL). Exploratory endpoints include biomarker analyses such as single-cell sequencing.

DETAILED DESCRIPTION:
This clinical trial is designed to evaluate the preliminary efficacy and safety of an oncolytic virus combined with chemotherapy and an immune checkpoint inhibitor in patients with initially unresectable, locally advanced esophageal squamous cell carcinoma (ESCC). The primary endpoints are safety, surgical conversion rate and event-free survival (EFS). Secondary endpoints include overall survival (OS), objective response r ate (ORR), and quality of life (QoL). Exploratory endpoints include biomarker analyses such as single-cell sequencing.

**Participant Procedures**:

1.All participants must undergo diagnostic endoscopy at West China Hospital to confirm eligibility. 2.Participants will undergo eligibility assessments. Once eligibility is confirmed, written informed consent will be obtained. 3.Single-cell sequencing of primary tumors or metastatic lymph nodes will be performed. All study-related costs will be covered by the research budget. 4.Participants will receive two to four cycles of the investigational treatment regimen (oncolytic virus + chemotherapy + PD-1 inhibitor), with each cycle lasting 21 days. Upon completion, patients will enter routine follow-up with healthcare professionals to monitor long-term safety and health status.

ELIGIBILITY:
Inclusion Criteria:

* A. Age 18-80 years B. Diagnosed with locally advanced esophageal squamous cell carcinoma (ESCC) with/without cervical lymph node metastases.

C. Ability to provide fresh tumor tissue samples (baseline) D. Normal major organ function E. Performance status (PS) score ≤ 1 F. Patients of childbearing potential must use contraception G. Voluntary participation with signed informed consent H. Able to comply with the study protocol, follow-up schedule, and other protocol requirements.

Exclusion Criteria:

* A. Received prior antitumor chemotherapy, radiotherapy, or immunotherapy before the first-line treatment.

B. High risk of gastrointestinal bleeding, esophageal fistula, or esophageal perforation C. Poor nutritional status D. Immune-related adverse events during prior radical treatment, such as Grade ≥3 pneumonitis, myocarditis, etc.

E. Signs and symptoms of interstitial diseases F. Presence of any severe and/or uncontrolled medical conditions G. Presence of concurrent malignancies H. Presence of other autoimmune diseases, or prolonged use of immunosuppressants or steroids I. Difficulty in patient communication or inability to comply with long-term follow-up J. Other conditions deemed unsuitable by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse effects (TRAEs) | Through study completion, an average of 1.5 year
  This study will collected any adverse medical events that occurred during the study drug treatment, and the treatment-related adverse events as assessed by CTCAE v5.0.
Event Free Survival (EFS) | Through study completion, an average of 1.5 year
  Time from the start of treatment to the first occurrence of any of the following events: disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | 24months
  Time from the start of treatment to death from any cause.
Objective Response Rate （ORR） | 12months
  The Objective Response Rate (ORR) is defined as the proportion of patients with complete response (CR) or partial response (PR), as assessed by RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No